CLINICAL TRIAL: NCT05133271
Title: Assessment of the Value of Passive Leg Raising (PLR) in Predicting the Onset of Maternal Arterial Hypotension and Norepinephrine Requirements After Spinal Anesthesia for Scheduled Cesarean Section.
Brief Title: Prediction of Maternal Arterial Hypotension After Spinal Anesthesia by Passive Leg Raise Test.
Acronym: EDLIDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210937; 2021-A01099-32 (Other: ID-RCB Number)
Record Dates: First submitted 2021-11-15; First posted 2021-11-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cesarean; Spinal Anesthesia
Keywords: Passive leg raise test (PLR); Cesarean section; Spinal anesthesia; Maternal arterial hypotension; Phenylephrine requirements; Norepinephrine requirements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Scheduled cesarean section (Experimental): Patient with scheduled cesarean section under spinal anesthesia.
  Interventions: Other: Clinical hemodynamic and echocardiographic evaluation

INTERVENTIONS:
Other: Clinical hemodynamic and echocardiographic evaluation — Clinical hemodynamic and echocardiographic evaluation in two stages T1 and T2, before performing the spinal anesthesia, carried out by a doctor different from the doctor in charge of the parturient in the operating room to ensure the blind hemodynamic results before the spinal anesthesia, in particular those of the passive leg raise test (PLR) :
  1. T1: clinico-echographic evaluation in dorsal decubitus position (45 °) with cushion under the right buttock.
  2. T2: clinico-ultrasound evaluation after performing the PLR.
     Then, clinical hemodynamic evaluation during two periods T3 and T4:
  3. T3: conditioning time of the parturient in the operating room during which clinical hemodynamic monitoring is set up and the basic values of arterial pressures (systolic, diastolic and mean) and heart rate are defined.
  4. T4: period after performing spinal anesthesia until clamping of the umbilical cord.

SUMMARY:
Spinal anesthesia for cesarean section is associated with a high incidence of low blood pressure. However, the pathophysiology of this arterial hypotension is not unequivocal and could involve, in addition to drug vasoplegia, a mechanical cause linked to lower caval compression or even true or relative hypovolemia. Passive leg raise test has been proposed in an attempt to identify parturients who are more likely to develop low blood pressure after spinal anesthesia. Nevertheless, the data available on this volume expansion test to predict hemodynamic variations after performing spinal anesthesia are still limited and few objective criteria have been described to predict this arterial hypotension.

The objective of the research is to study the hypothesis according to which the presence of hypovolaemia (true or relative) objectified by a positive passive leg raise test would cause hypotension more frequent and more marked in intensity.

DETAILED DESCRIPTION:
Spinal anesthesia for cesarean section is associated with a high incidence of low blood pressure. However, the pathophysiology of this arterial hypotension is not unequivocal and could involve, in addition to drug vasoplegia, a mechanical cause linked to lower caval compression or even true or relative hypovolemia.

Passive leg raise test has been proposed in an attempt to identify parturients who are more likely to develop low blood pressure after spinal anesthesia. Nevertheless, the data available on this volume expansion test to predict hemodynamic variations after performing spinal anesthesia are still limited and few objective criteria have been described to predict this arterial hypotension.

The objective of the research is to study the hypothesis according to which the presence of hypovolaemia (true or relative) objectified by a positive passive leg raise test would cause hypotension more frequent and more marked in intensity.

Patients will have a clinical hemodynamic and echocardiographic evaluation, before performing the spinal anesthesia, before and after the passive leg raise test.

Then, the patients will benefit from a clinical hemodynamic evaluation during the preparation of the parturient in the operating room and finally after the completion of the spinal anesthesia and until the clamping of the umbilical cord.

ELIGIBILITY:
Inclusion Criteria:

* Adult women admitted to Necker Enfants Malades hospital for scheduled cesarean section under spinal anesthesia
* Written informed consent

Exclusion Criteria:

* No health insurance
* Urgent cesarean
* Failure of spinal anesthesia
* Free and informed consent impossible to obtain (especially due to a language barrier)
* Severe cardiovascular or neurovascular comorbidities
* Contraindication to the PLR (intracranial hypertension, fractures of the pelvis and / or lower limbs, ...)
* Background of preeclampsia or eclampsia
* Severe fetal pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient with scheduled cesarean section under spinal anesthesia.
Enrollment: 64 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
Maternal arterial hypotension | Day 0
  Maternal arterial hypotension following spinal anesthesia. Maternal hypotension is defined as a drop in systolic blood pressure (SBP)> 20% of baseline.
Positivity of passive leg raise test | Day 0
  A positive passive leg raise test is defined as an increase in the Subaortic Flow Velocity Time Integral of 10% or more. The increase in cardiac output is measured by a cardiac ultrasound.
Positive passive leg raise test performance | Day 0
  Performance of a positive passive leg raise test in predicting the onset of maternal arterial hypotension after spinal anesthesia. Significant performance will be defined by sensitivity and specificity > 90%.

SECONDARY OUTCOMES:
Total dose of norepinephrine | Day 0
  Total dose of norepinephrine received during the procedure from the beginning of the spinal anesthesia injection up to umbilical cord clamping measured in micrograms.
Onset of severe arterial hypotension | Day 0
  Onset of severe arterial hypotension defined as a drop in systolic blood pressure greater than 30% of baseline.
Onset of nausea and vomiting | Day 0
  Onset of nausea and vomiting from the spinal anesthesia injection up to the end of the c-section.
Occurrence of disturbances of consciousness | Day 0
  Occurrence of consciousness alteration assessed by the Glasgow Coma Scale (from Teasdale G & Jennett B. Lancet 1974).
  Three aspects of behavior are measured independently: motor response, verbal response and eye opening.
  Each component has a number of grades starting with the most severe. The best ocular response has 4 grades; the best verbal response has 5 grades; the best motor response has 6 grades.
  Rating: the score of each component as well as the sum of the components are considered. The total score is out of 15 points; lower scores indicating more severe impairment. The lowest possible score is 3, indicating deep coma or death, and the highest possible score is 15, indicating a fully awake individual.
Occurrence of sedation and agitation | Day 0
  Occurrence of sedation and agitation during the c-section assessed by the Richmond Agitation-Sedation scale (RASS).
  This score is based on the observation of the patient It has 10 stages ranging from +4 (combative patient) to -5 (patient who cannot be woken up).
Assessment of fetal well-being | Day 0
  Evaluation of fetal well-being by fetal heartbeat, by the Apgar score at 1, 3 and 5 minutes of life, and study of the pH in the umbilical cord, a pH value <7.2 defines fetal distress.
Quality of ultrasound images | Day 0
  Assessment of obtaining views (parasternal long-axis view, parasternal short-axis view, apical 4-chamber view, subcostal).
  Interpretability of the measurements obtained.
Relative or absolute hypovolemia | Day 0
  Describe the echocardiographic parameters reflecting the different physiopathological mechanisms at the origin of arterial hypotension secondary to spinal anesthesia of the parturient at the end of pregnancy.
  To note the parameters suggestive of relative or absolute hypovolaemia: inferior vena cava diameter < 8 mm; "kissing sign" of the left ventricle, defined as à end-systolic collapse of the left ventricle; E/A ratio < 1.
Right ventricle systolic or diastolic dysfunction | Day 0
  Describe the echocardiographic parameters reflecting the different physiopathological mechanisms at the origin of arterial hypotension secondary to spinal anesthesia of the parturient at the end of pregnancy.
  Right ventricle systolic function: measurement of the TAPSE (tricuspid annular plane systolic excursion; presence of a paradoxical septal motion (yes/no).
  Right ventricle diastolic function: presence of right ventricle dilation defined as end-diastolic right ventricle area (EDRVA) / end-diastolic left ventricle area (EDLVA) > 0.6; "severe" dilatation is defined as a ratio > 1.
Left ventricle systolic and diastolic dysfunction | Day 0
  Describe the echocardiographic parameters reflecting the different physiopathological mechanisms at the origin of arterial hypotension secondary to spinal anesthesia of the parturient at the end of pregnancy.
  Left ventricle systolic function:
  left ventricle ejection fraction (LVEF) - apical-4-chamber view - defined as LVEF = (EDLVA-ESLVA)/EDLVA Left ventricle shortening fraction (LVSF) - parasternal short-axis view - defined as LVSF = (EDLVA-ESLVA)/EDLVA MAPSE (mitral annular plane systolic excursion
  Left ventricle diastolic function:
  Mitral flow profile: E wave / A wave ratio Left atrium area (cm²)
Pericardial effusion | Day 0
  Describe the echocardiographic parameters reflecting the different physiopathological mechanisms at the origin of arterial hypotension secondary to spinal anesthesia of the parturient at the end of pregnancy.
  Measurement of the size (in mm) of the pericardial effusion (left and right ventricles lateral walls).
Maternal comfort during the passive leg raising | Day 0
  Assessment of the maternal comfort during the passive leg raising test with a numerical scale (from 0: maximal discomfort to 10: maximal comfort).
Heart rate | Day 0
  Association of increased up heart rate and total dose of neosynephrine at the end of the c-section.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Repessé, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Hawa Keita-Meyer, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No